CLINICAL TRIAL: NCT01990950
Title: Evaluation of the Long-term Safety and Performance of the Zenith® Fenestrated Abdominal Aortic Aneurysm (AAA) Endovascular Graft Post-Approval Study
Brief Title: Fenestrated AAA Endovascular Graft Post-Approval Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-005
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Results first posted 2021-09-14 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Abdominal Aortic Aneurysm (AAA); Aorto-iliac Aneurysm; Juxtarenal Aneurysm
Keywords: Aneurysm; Aortic Aneurysm; Iliac Aneurysm; Aortic Aneurysm, Abdominal; Vascular Diseases; Cardiovascular Diseases; Aortic Diseases
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm; Aortic Aneurysm; Iliac Aneurysm; Vascular Diseases; Cardiovascular Diseases; Aortic Diseases

ARMS (1):
- Zenith® Fenestrated AAA Endovascular Graft (Experimental)
  Interventions: Device: Zenith® Fenestrated AAA Endovascular Graft

INTERVENTIONS:
Device: Zenith® Fenestrated AAA Endovascular Graft — The Zenith® Fenestrated AAA Endovascular Graft with the H&L-B One-Shot™ Introduction System is indicated for the endovascular treatment of patients with abdominal aortic or aortoiliac aneursyms having morphology suitable for endovascular repair

SUMMARY:
This post-market study is approved by the US FDA to evaluate the long-term safety and performance of the Zenith® Fenestrated AAA Endovascular Graft.

ELIGIBILITY:
Inclusion Criteria:

* abdominal aortic and aortoiliac aneursyms with a diameter greater than or equal to 5 cm
* aortic or aortoiliac aneurysm with a history of growth greater than or equal to 0.5 cm per year, or clinical indication for AAA repair

Exclusion Criteria:

* proximal neck less than 4mm or greater than or equal to 15 mm in length unless otherwise compromised to preclude seal
* renal artery stenosis greater than 50 percent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-03; Primary Completion 2020-10-12 (Actual); Study Completion 2020-10-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of California-Davis, Sacramento, California
  - University of Colorado, Aurora, Colorado
  - Borgess Research Institute, Kalamazoo, Michigan
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Wake Forest University Health, Winston-Salem, North Carolina
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zenith® Fenestrated AAA Endovascular Graft
Started | 21
Completed | 10
Not Completed | 11
Not completed — Death | 3
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Groups:
- Zenith® Fenestrated AAA Endovascular Graft: The Zenith® Fenestrated AAA Endovascular Graft is a modular system consisting of three components, a proximal body graft, a distal bifurcated body graft and one iliac leg. Additional ancillary components (main body extensions, iliac leg extensions, converters, and occluders) are available. The Zenith® Alignment Stent is a balloon-expandable stent that can be deployed through scallops or fenestrations in a Zenith® Fenestrated AAA Endovascular Graft into branch vessels of the aorta.
Arm/Group | Zenith® Fenestrated AAA Endovascular Graft
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  White | 19
  White; Hispanic or Latino | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Treatment Success : AAA Related Mortality
Description: patients treated with the Zenith® Fenestrated AAA Endovascular Graft will have a rate of aneurysm-related mortality at 5 years that meets a performance goal of 18% ,
Time Frame: 5 years
Population: patients with abdominal aortic or aortoiliac aneurysms having morphology suitable for endovascular repair
Measure: Count of Participants; unit: Participants
Arm/Group | Zenith® Fenestrated AAA Endovascular Graft
Number analyzed (Participants) | 21
Participants | 0

ADVERSE EVENTS:
Time Frame: 5 years
Groups:
- Zenith® Fenestrated AAA Endovascular Graft: The Zenith® Fenestrated AAA Endovascular Graft is a modular system consisting of three components, a proximal body graft, a distal bifurcated body graft and one iliac leg.
Arm/Group | Zenith® Fenestrated AAA Endovascular Graft
All-Cause Mortality (participants affected / at risk) | 3/21
Serious Adverse Events (participants affected / at risk) | 11/21
Other Adverse Events (participants affected / at risk) | 13/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zenith® Fenestrated AAA Endovascular Graft (N=21)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (4)
Atrial flutter (Cardiac disorders) | 1 (2)
Atrioventricular block second degree (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 3 (3)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1)
Stent-graft endoleak (General disorders) | 2 (3)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Gallbladder mass (Hepatobiliary disorders) | 1 (1)
Biliary tract infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1)
Dialysis (Surgical and medical procedures) | 1 (1)
Transfusion (Surgical and medical procedures) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zenith® Fenestrated AAA Endovascular Graft (N=21)
Atrial fibrillation (Cardiac disorders) | 2 (5)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (4)
Stent-graft endoleak (General disorders) | 2 (3)
Pneumonia (Infections and infestations) | 2 (2)
Transfusion (Surgical and medical procedures) | 2 (2)
Aortic aneurysm (Vascular disorders) | 3 (3)
Renal infarct (Renal and urinary disorders) | 3 (3)
Myocardial ischaemia (Cardiac disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/50/NCT01990950/Prot_000.pdf